CLINICAL TRIAL: NCT04180969
Title: Impact of Repetitive Transcranial Magnetic Stimulation (rTMS) of Limbic Brain Circuitry in Stress Modulation in a Healthy Population
Brief Title: rTMS of Limbic Circuitry in Stress Modulation in Healthy Volunteers
Acronym: TSM-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: TSM-1
Record Dates: First submitted 2019-11-24; First posted 2019-11-29 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Stress; Healthy
MeSH Terms: interventions — Yohimbine; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Double-blind, 1Hz mPFC (vs. sham) rTMS X stressor (vs. placebo), 4-session, within-subjects, randomized crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: sham (inactive) figure of 8 coil for rTMS, and placebo for pharmacological stressor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo stressor, sham rTMS (Placebo Comparator): placebo stressor is lactose, and sham rTMS is inactive figure of 8 coil
  Interventions: Drug: Placebo oral tablet; Device: sham rTMS
- placebo stressor, active rTMS (Experimental): placebo stressor is lactose, and active rTMS is 1Hz stimulation over the medial prefrontal cortex
  Interventions: Device: medial prefrontal cortex rTMS; Drug: Placebo oral tablet
- active stress, sham rTMS (Experimental): active stressor is the combination of yohimbine 54mg + hydrocortisone 20mg, and sham rTMS is inactive figure of 8 coil
  Interventions: Drug: yohimbine + hydrocortisone; Device: sham rTMS
- active stress, active rTMS (Experimental): active stressor is the combination of yohimbine 54mg + hydrocortisone 20mg, and active rTMS is 1Hz stimulation over the medial prefrontal cortex
  Interventions: Drug: yohimbine + hydrocortisone; Device: medial prefrontal cortex rTMS

INTERVENTIONS:
Drug: yohimbine + hydrocortisone — yohimbine 54mg + hydrocortisone 20mg oral
  Arms: active stress, active rTMS; active stress, sham rTMS
Device: medial prefrontal cortex rTMS — 1 Hz mPFC rTMS
  Arms: active stress, active rTMS; placebo stressor, active rTMS
Drug: Placebo oral tablet — placebo stressor
  Arms: placebo stressor, active rTMS; placebo stressor, sham rTMS
Device: sham rTMS — sham mPFC rTMS
  Arms: active stress, sham rTMS; placebo stressor, sham rTMS

SUMMARY:
This study will be conducted with healthy male and female participants. Aim 1 will determine during sham repetitive transcranial magnetic stimulation (rTMS) how a drug stressor combination (yohimbine + hydrocortisone) relative to placebo alters : (1a) impulsivity; (1b) mood; and (1c) physiology. Aim 2 will determine whether active rTMS over the medial prefrontal cortex alters the effects of stress-exposure on (2a) decision-making, (2b) mood, and (2c) biomarkers of stress.

DETAILED DESCRIPTION:
This study will use a double-blind, within-subjects randomized crossover design. Each participant will complete 4 sessions in this two-factor (2x2) combinatorial design: 1Hz medial prefrontal cortex (mPFC) vs. sham repetitive transcranial magnetic stimulation (rTMS) X pharmacological stressor (yohimbine 54mg + hydrocortisone 20mg) vs. placebo, with each session separated by at least 1 week. Participants will be asked not to use alcohol or drugs for 24-hr before arriving at the lab. We expect to complete screen at least 20 individuals to complete 12 individuals in this study. Candidates will first undergo psychiatric and medical screening to rule out contraindications to participation. Once enrolled, each participant will complete, in randomized order, the 4 conditions above. Periodic measures will be collected before and after the rTMS/sham and stress/placebo interventions. These measures will include subjective, behavioral and physiological assessments, as well as saliva and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60 yr
* Right-handed
* Males and non-pregnant/non-lactating females
* Cognitively intact (total IQ score >80 on Shipley Institute of Living Scale)
* Screening cardiovascular indices must be within ranges that allow for safe use of stressor: resting HR 50-90 bpm, systolic BP 90-140 mmHg, and diastolic BP 50-90 mmHg
* Use alcohol and/or marijuana <3 times/week; each "time" should consist of <1 marijuana "joint" equivalent and <3 alcoholic drinks

Exclusion Criteria:

* Under influence of any substance during session
* Past 7-day use of illicit drugs (excluding marijuana) based on Timeline Followback interview
* Urine positive for opioids, cocaine metabolites, benzodiazepines, barbiturates, amphetamines or pregnancy
* Medical conditions prohibiting use of rTMS (e.g. seizure history; using validated rTMS screening instrument)
* Lifetime diagnosis of: psychotic disorder, bipolar disorder, generalized anxiety disorder, obsessive compulsive disorder, or major depression that is not substance-induced
* Past-year substance use disorder
* Medical conditions making it unsafe for participation (e.g. neurological, cardiovascular, pulmonary, or systemic diseases)
* Lactose intolerance (placebo dose)
* Any prohibited medications: medications that lower seizure threshold, psychiatric medications, prescription pain medications, or blood pressure medications
* Chronic head or neck pain
* Taken part in any research studies in the past month

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Color-Word Stroop Task | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  reaction time (msec) measure of cognitive interference
Digit Span Task | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  number of digits recalled, measure of verbal working memory
Wisconsin Card Sorting Task | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  number of correct items, measure of ability to shift set and assesses cognitive flexibility
Monetary Incentive Delay Task | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  number of rewards received, measure of motivation
Delay Discounting Task | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  rate of monetary discounting
Effort Choice Task | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  number of progressive ratio (PR) choices vs. fixed ratio (FR) choices
Positive and Negative Affect Schedule (PANAS) positive affect | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  10-item questionnaire sub scale that measures positive affect
Positive and Negative Affect Schedule (PANAS) negative affect | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  10-item questionnaire sub scale that measures negative affect
State-Trait Anxiety Inventory | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  questionnaire subscale that measures state anxiety
Blood pressure | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  Blood pressure (mm Hg)
Heart rate | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  Heart rate (beats/min)
Saliva cortisol level | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  Saliva cortisol level (µg/mL)
Saliva alpha-amylase level | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  Saliva alpha-amylase level (U/mL)
Plasma prolactin level | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  Plasma prolactin level (pg/mL)
Plasma BDNF level | change from pre- to post-intervention in each of the 4 sessions (through study completion, about 1 month total)
  Plasma brain derived neurotrophic factor level (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Greenwald, PhD, Study Director — Wayne State University

IPD SHARING:
Plan to Share IPD: Yes
Full sharing plan is being developed.
Supporting Information: Study Protocol
Time Frame: Materials will only become available after the study is completed and the first manuscript from this project is published.
Access Criteria: Qualified investigators may apply in writing to Dr. Greenwald